CLINICAL TRIAL: NCT02797613
Title: Restricted Reporting for Positive Urine Cultures Randomized Controlled Trial
Brief Title: Restricted Reporting for Positive Urine Cultures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial University of Newfoundland (Other)
Responsible Party: Principal Investigator, Peter Daley, Assistant Professor, Memorial University of Newfoundland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MUN-01
Record Dates: First submitted 2016-06-08; First posted 2016-06-13 (Estimated); Results first posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Bacteriuria; Urinary Tract Infection
MeSH Terms: conditions — Bacteriuria; Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restricted Reporting (Experimental): Microbiology laboratory will report "Positive urine cultures may represent asymptomatic bacteriuria or urinary tract infection. If urinary tract infection is suspected clinically, please call 777-xxxx (researcher mobile phone) for identification and susceptibility results"
  Interventions: Behavioral: Restricted Reporting
- Standard Reporting (No Intervention): Microbiology laboratory will report identification and susceptibility results

INTERVENTIONS:
Behavioral: Restricted Reporting — An abbreviated version of the microbiology report indicating that growth is present and the physician should call the lab for further details if clinically important
  Arms: Restricted Reporting

SUMMARY:
Asymptomatic bacteriuria (AB) is a condition in which bacteria are detected in urine culture without urinary symptoms. The inappropriate use of antibiotic treatment for AB selects bacterial flora to express resistance mutations. Reducing inappropriate antibiotic use for AB is difficult, since the microbiology laboratory cannot distinguish patients with AB. The investigators study will use a restricted laboratory report requesting the physician to call the laboratory for culture results. The restricted report may reduce the rate of inappropriate treatment of AB.

DETAILED DESCRIPTION:
Positive urine cultures during the study period will be randomized to restricted microbiology laboratory reporting or standard microbiology laboratory reporting. Physician or patient consent will not be collected. Patient records will be assessed by the investigator to determine if patients have AB or urinary tract infection. Physician antibiotic treatment decision in both groups will be collected.

ELIGIBILITY:
Inclusion Criteria:

* positive urine culture from inpatients at Health Sciences Centre or St. Clare's Mercy Hospital or outpatients during study period.

Exclusion Criteria:

* pregnancy,
* antibiotic treatment at the time of urine collection,
* collection from an indwelling catheter,
* admission to long term care facility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Daley, MD FRCPC, Principal Investigator — Memorial University
Locations (1):
- Health Sciences Center, St. John's, Newfoundland and Labrador, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Daley P, Garcia D, Inayatullah R, Penney C, Boyd S. Modified Reporting of Positive Urine Cultures to Reduce Inappropriate Treatment of Asymptomatic Bacteriuria Among Nonpregnant, Noncatheterized Inpatients: A Randomized Controlled Trial. Infect Control Hosp Epidemiol. 2018 Jul;39(7):814-819. doi: 10.1017/ice.2018.100. Epub 2018 May 28. PMID 29804552

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Restricted Reporting | Standard Reporting
Started | 55 | 55
Completed | 55 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 110 Results randomized. All randomized results were analysed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Restricted Reporting | Standard Reporting | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (16.3) | 68.6 (16.0) | 68.1 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 36 | 71
  Male | 20 | 19 | 39
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 55 | 55 | 110
Asymptomatic Bacteriuria [Count of Participants; unit: Participants] | 35 | 41 | 76

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients Receiving Appropriate Treatment
Description: Sum of urinary tract infection treated and asymptomatic bacteriuria not treated
Time Frame: 72 hours from positive culture
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Restricted Reporting | Standard Reporting
Number analyzed (Participants) | 55 | 55
Participants | 44 | 29

ADVERSE EVENTS:
Time Frame: 7 days after positive urine culture
Description: Bacteremia and Death reported at 7 days follow up, Adverse events (systemic inflammatory response syndrome) reported at 72 hours follow up
Arm/Group | Restricted Reporting | Standard Reporting
All-Cause Mortality (participants affected / at risk) | 2/55 | 1/55
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 7/55 | 9/55
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Restricted Reporting (N=55) | Standard Reporting (N=55)
Bacteremia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) — 7 days after positive urine culture
Tachycardia (Cardiac disorders) | 4 (4) | 5 (5)
Edema (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Abnormal Body Temperature (General disorders) | 0 (0) | 0 (0)
Hyperglycaemia (Endocrine disorders) | 0 (0) | 0 (0)
Elevated White Blood Cell Count (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Altered Mental Status (Nervous system disorders) | 2 (2) | 5 (5)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
Our design is a proof-of-concept which will require additional trials to verify. It would be impractical to manually screen all inpatient urine specimens using our inclusion criteria, although automated eligibility screening may be possible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-26): https://cdn.clinicaltrials.gov/large-docs/13/NCT02797613/Prot_SAP_000.pdf